CLINICAL TRIAL: NCT00111527
Title: An Assessment of the Echo-guided Optimal Cardiac Resynchronization Therapy in Patients Undergoing 'Ablate And Pace' Therapy for Permanent Atrial Fibrillation
Brief Title: APAF: Assessment of Cardiac Resynchronization Therapy in Patients With Permanent Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1893A
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2025-06-12 (Actual); Status verified 2010-03

CONDITIONS: Congestive Heart Failure; Atrial Fibrillation
Keywords: Heart failure; Atrial fibrillation; Cardiac resynchronization; Cardiac pacing; Catheter ablation; Quality of life; Echocardiography
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Normal RV pacing
  Interventions: Other: normal RV pacing
- 2 (Experimental): Echo-guided optimization of pacing
  Interventions: Other: Optimized echo-guided CRT pacing

INTERVENTIONS:
Other: Optimized echo-guided CRT pacing — Echo-TDI guided VV-delay optimization
  Arms: 2
Other: normal RV pacing — PM or ICD implant according to patient indication
  Arms: 1

SUMMARY:
A suboptimal level of resynchronization (cardiac resynchronization therapy [CRT]) achieved in many patients with actual standards and techniques based on tissue-Doppler echocardiography could be more effective to obtain better CRT results. Eligible patients who successfully received atrioventricular (AV) junction ablation and biventricular (BiV) pacing are randomised to a comparison between a strategy of right ventricular (RV) apical pacing with delayed CRT based on clinical indications with a strategy of early optimal CRT based on an echocardiographic stratification.

End-points:

* Acute echo comparison (acute echo study)
* Quality of life and exercise tolerance (Short-term clinical study)
* Composite end-point of CRT clinical failure (Long-term clinical study)

DETAILED DESCRIPTION:
Background: Cardiac resynchronization therapy (CRT) in patients in atrial fibrillation (AF) seems to provide modest favorable effect compared with RV pacing. In the Optimal Pacing SITE (OPSITE) trial the results were heterogeneous. The situation was almost certainly one in which some patients are showing marked clinical benefit with LV-based pacing, balanced by other patients in whom RV was the best choice. Therefore with the actual standards, CRT pacing cannot be recommended as a first line treatment for all patients with AF and refractory heart failure and new criteria to identify the patients who might benefit are needed. Furthermore, a pre-requisite for CRT in patients with AF is the presence of stable 3rd degree AV block which usually implies the need for performing catheter ablation of the AV junction.

Study hypothesis: We hypothesized that a suboptimal level of resynchronization is achieved in many patients with actual standards and that some techniques based on tissue-Doppler echocardiography could be more effective to obtain better (hopefully optimal) CRT results.

Objective: The aim of the APAF+ heart failure (HF) trial is to compare, in patients affected by permanent AF and refractory heart failure, a strategy of delayed CRT based on clinical indications with a strategy of early optimal CRT based on an echocardiographic stratification.

Study protocol: Eligible patients who successfully received AV junction ablation and biventricular pacing are randomised to a comparison between a strategy of RV apical pacing with delayed CRT based on clinical indications with a strategy of early optimal CRT based on an echocardiographic stratification. The optimal CRT is defined as the shortest intra-LV delay obtained with tissue-doppler echocardiography among RV, LV and BiV optimised VV interval.

An acute echocardiographic evaluation is performed shortly after randomisation. A short-term clinical evaluation is performed after 6 months. A long-term clinical evaluation is performed up to 24 months.

End-points:

* Acute echo comparison (acute echo study)
* Quality of life and exercise tolerance (Short-term clinical study)
* Composite end-point of CRT clinical failure (Long-term clinical study)

Study size: The study will randomise 458 patients and will be conducted in 46 centres with an average of 10 patients per centre. Patient enrolment time is anticipated to last 2 years. As the study will continue for a period of 12 months after the enrolment of the last patient, total study duration will be approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with permanent AF in whom a clinical decision had been made to undertake complete AV junction ablation and ventricular pacing because of drug-refractory, severely symptomatic, uncontrolled high ventricular rate
* Patients with permanent AF, drug-refractory heart failure, depressed LV function in whom a clinical decision had been made to undertake left ventricular synchronization pacing

Exclusion Criteria:

* New York Heart Association class IV heart failure, or systolic blood pressure ≥80 mmHg
* Severe concomitant non cardiac disease
* Need for surgical intervention
* Myocardial infarction within 3 months
* Primary hypertrophic cardiomyopathy
* Arrhythmogenic right ventricular dysplasia
* Primary valvular heart disease
* Sustained ventricular tachycardia or ventricular fibrillation
* Previously implanted pacemaker
* Inability to obtain reliable RV and LV pacing and persistent AV block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2005-05; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Short-term clinical study (6 months): Quality of life (measured as Minnesota Living with Heart Failure Questionnaire, Specific Symptom Scale and New York Heart Association classification) and exercise capacity at 6 months in the 2 study groups | 6 months
Long-term clinical study (24 months): Composite end-point of: death due to cardiovascular cause, hospitalisation for worsening heart failure, worsening heart failure or failure to achieve a persistent subjective symptom improvement (clinical failure) | 24 months

SECONDARY OUTCOMES:
The evaluation of the predictive value of echo desynchronisation indexes (inter and intra-LV delays) for identification of clinical failure (see above) | 24 months
Cost-benefit comparison of the 2 pacing strategies | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Brignole, MD, Principal Investigator — Ospedali del Tigullio, Lavagna, Italy; Carlo Menozzi, MD, Principal Investigator — Ospedale S Maria Nuova, Reggio Emilia, Italy
Locations (2):
- Italy (2):
  - Michele Brignole, Lavagna, Genova
  - Arcispedale S Maria Nuova, Reggio Emilia, Reggio Emilia

REFERENCES:
- [Background] Brignole M, Gammage M, Puggioni E, Alboni P, Raviele A, Sutton R, Vardas P, Bongiorni MG, Bergfeldt L, Menozzi C, Musso G; Optimal Pacing SITE (OPSITE) Study Investigators. Comparative assessment of right, left, and biventricular pacing in patients with permanent atrial fibrillation. Eur Heart J. 2005 Apr;26(7):712-22. doi: 10.1093/eurheartj/ehi069. Epub 2004 Dec 20. PMID 15618036
- [Background] Wood MA, Brown-Mahoney C, Kay GN, Ellenbogen KA. Clinical outcomes after ablation and pacing therapy for atrial fibrillation : a meta-analysis. Circulation. 2000 Mar 14;101(10):1138-44. doi: 10.1161/01.cir.101.10.1138. PMID 10715260
- [Background] Auricchio A, Abraham WT. Cardiac resynchronization therapy: current state of the art: cost versus benefit. Circulation. 2004 Jan 27;109(3):300-7. doi: 10.1161/01.CIR.0000115583.20268.E1. No abstract available. PMID 14744954
- [Derived] Brignole M, Botto G, Mont L, Iacopino S, De Marchi G, Oddone D, Luzi M, Tolosana JM, Navazio A, Menozzi C. Cardiac resynchronization therapy in patients undergoing atrioventricular junction ablation for permanent atrial fibrillation: a randomized trial. Eur Heart J. 2011 Oct;32(19):2420-9. doi: 10.1093/eurheartj/ehr162. Epub 2011 May 23. PMID 21606084